CLINICAL TRIAL: NCT03500770
Title: Transcranial Direct Current Stimulation (tDCS) for Cognitive Deficit, Fatigue and Pain in Patients With Post Treatment Lyme Disease Syndrome
Brief Title: Lyme Disease Patients With Memory Problems
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Nevena Zubcevik, Attending Physcian/Instructor, Department of Physical Medicine and Rehabilitation, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P000309
Record Dates: First submitted 2016-10-13; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Lyme Disease
Keywords: Post Treatment Lyme Disease Syndrome
MeSH Terms: conditions — Lyme Disease; Post-Lyme Disease Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial Direct Current Stimulator (Experimental): The Transcranial Direct Current Stimulator device (tDCS) is a safe technique which poses a non-significant risk to study subjects. This technique uses weak current which is applied by using two electrodes. In the literature, no undesirable or long-lasting side effects due to device have been reported, nor have any participants reportedly abandoned a study due to discomfort.
  Interventions: Device: Transcranial Direct Current Stimulator

INTERVENTIONS:
Device: Transcranial Direct Current Stimulator — The tDCS device to be used will be an investigational, battery powered, custom-made stimulator able to deliver a biphasic alternate current. Active stimulation consists of 10 active tDCS sessions with current intensity fixed at 2mA for 20 minutes. It has been safely used in several other research studies. The side effects profile for this type of stimulation include tingling/itching at the site of stimulation, skin irritation/redness at the site of stimulation, headache or dizziness.

SUMMARY:
The main purpose of this study is to see if a device known as Transcranial Direct Current Stimulator (tDCS) is helpful in reducing persistent symptoms after Lyme disease treatment. Some of these symptoms include problems with memory, fatigue or pain.

DETAILED DESCRIPTION:
Lyme disease is a tick-borne illness caused by Borrellia Bugdorferi after tick bite. This disease mostly presents with a skin rash which looks like bulls eye and therefore known as bulls-eye skin rash or Erythema Migrans. The standard of care of Lyme disease is a few weeks of antibiotics. Most of the patients do well after antibiotics treatment. However 10-20% of patients go on to develop persistent symptoms such as memory problems, fatigue and pain several months after the antibiotics treatment. Such symptoms are collectively known as Post Treatment Lyme Disease Syndrome. In this study we want to see if a device known as Transcranial Direct Current Stimulator (tDCS) is helpful in reducing these symptoms after Lyme disease treatment.

This study will consist of a total of 13 visits. After determining eligibility criteria through pre-screening and labs we will schedule visit 1. During visit 1 we will ask the study participants to fill several questionnaire forms related to memory, pain, fatigue, quality of life, depression and headache etc. We will draw blood to measure certain lab markers. We will do a few other tests to determine brain oxygenation level and to check brain waves.

During next 10 visits we will administer small current through a device known as Transcranial Direct Current Stimulator. This device and the amount of current delivered is very safe. Visit 12 is fairly the same as visit 1 as we will ask the study participant to answer questions related to memory, quality of life, pain, fatigue, depression and headache. During this visit we will also do the test to determine oxygenation level of brain and will perform brain wave testing.

Visit 13 will be last and final visit which will occur one month after visit 12. During this final visit the study participant will be asked to answer the questions related to memory, quality of life, pain, fatigue, depression and headache. During this visit we will again measure oxygenation level of brain and perform brain wave testing.

By doing this study in total 13 visits we expect to find out if the device "Transcranial Direct Current Stimulator" is helpful in reducing these symptoms after Lyme disease treatment.

ELIGIBILITY:
Fifteen subjects will be selected to take part in this study. All subjects must meet the following criteria:

* Inclusion criteria:

  1. Age over 18 years, both males and females
  2. History of Lyme disease as diagnosed per CDC criteria and/or evidence of Erythema Migrans or diagnosis of Lyme disease as documented in medical record by an experienced health care practitioner.
  3. Meet defining criteria of Post Treatment Lyme Disease Syndrome (PTLDS) proposed by Infectious Diseases Society of America (IDSA)
  4. Ability to give informed consent as assessed by study physician
  5. Willing to participate in 10 tDCS sessions over two week period
  6. If on long-term antibiotics or supplements for treatment of Lyme disease must be willing to keep treatment regimen consistent during participation in the study
* Exclusion criteria:

  1. Evidence of any active Borrelia infection or co-infection such as Babesiois, Anaplasmosis, Erhlichiosis, Ricketsia as assessed by serum serology, such patient will be referred to ID
  2. Evidence of current or prior infection by B. Mioymoti or B. hemsii, such patients will be referred to ID
  3. Any of the exclusion criteria of Post Treatment Lyme Disease Syndrome (PTLDS) as proposed by Infectious Diseases Society of America (IDSA)
  4. History of other chronic inflammatory conditions such as:

     * Rheumatoid arthritis
     * Asthma
     * Autoimmune diseases
     * Chronic prostatitis
     * Glomerulonephritis
     * Celiac disease
     * Inflammatory bowel disease
     * Pelvic inflammatory disease
     * Interstitial cystitis
     * Vasculitis
  5. Existence of major neurologic or psychiatric condition such as epilepsy, severe depression or others
  6. Past history of neurosurgery
  7. History of significant alcohol or drug abuse during previous 6 months
  8. Presence of unstable medical conditions such as uncontrolled diabetes mellitus, cardiac pathology, cancer, kidney insufficiency, acute thrombosis or others
  9. Any new medication or dosage changes in the past 60 days interfering with your symptoms related to PTLDS
  10. Concurrent use of opioids or narcotics which cause CNS suppression, cognitive or motor slowing
  11. Concurrent use of muscle relaxants
  12. Concurrent use of anti-epileptics such as Carbamazepine
  13. Pregnancy as assessed by urine pregnancy test
  14. Contraindication to tDCS such as metal in the head or implanted electronic medical devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitive dysfunction | up to 12 weeks
  CVLT test change from baseline

SECONDARY OUTCOMES:
Fatigue | up to 12 weeks
  GSQ Questionnaire change from baseline

OTHER OUTCOMES:
Pain | up to 12 weeks
  Analog scale pain level change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nevena Zubcevik, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Nevena Zubcevik, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No